CLINICAL TRIAL: NCT03772132
Title: A Multicentre, Open-label, Randomised, Controlled Study of Molecularly Precision Target Therapy Based on Tumor Molecular Profiling With FORFIRINOX in Advanced or Recurrent Extrahepatic Cholangiocarcinoma and Gallbladder Carcinoma
Brief Title: Chemothetapy FORFIRINOX in Advanced or Recurrent Extrahepatic Cholangiocarcinoma and Gallbladder Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other); RenJi Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, liu yingbin, head of general surgery department，xin hua Hospital Affiliation: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLY20181206
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Cholangiocarcinoma of the Extrahepatic Bile Duct; Gallbladder Cancer
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Mutation

ARMS (1):
- Chemotherapy (Experimental): The patients wil receive conventional chemotherapy FORFIRINOX
  Interventions: Biological: mutation and signal pathway activation status analysis Drug: FORFIRINOX

INTERVENTIONS:
Biological: mutation and signal pathway activation status analysis Drug: FORFIRINOX — Conventional chemotherapy:5FU plus irinote- can plus oxaliplatin combination therapy

SUMMARY:
The purpose of this study is to evaluate the feasibility, efficacy and safety of FORFIRINOX in advanced or recurrent extrahepatic cholangiocarcinoma and gallbladder carcinoma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility, efficacy and safety of FORFIRINOX in advanced or recurrent extrahepatic cholangiocarcinoma and gallbladder carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* • Chinese；

  * Stable vital signs, KPS≥60;
  * Patients have a diagnosis of advanced or recurrent metastatic extrahepatic cholangiocarcinoma or gallbladder carcinoma by histopathology or cytopathology, who are not suitable for radical surgery or have progressed R1 resection or palliative surgery;
  * Adequate fresh tumor tissue for genome sequencing and immuno- histochemistry test; harboring mutations or abnormal activation of erb-b2 receptor tyrosine kinase signal pathway components;
  * At least one measurable and evaluable site of disease according to the RECIST criteria version 1.1;
  * Life expectancy of more than 12 weeks;
  * Adequate hepatic, hematologic and renal functions(ALT≤10×upper limit of normal (ULN), AST≤10×ULN, the Child-Pugh classification for class A or B, white blood cells≥3×10^9/L, neutrophils≥1.5×10^9/L, platelets≥80×10^9/L , hemoglobin ≥ 90g/L, creatinine clearance rate≥60ml/min;
  * Volunteer for this study, have written informed consent and have good Patient compliance;
  * Female patients of childbearing potential and their mates agree to avoid pregnancy.

Exclusion Criteria:

* Have received following treatment before this study:

  1. Anti-tumor molecular target therapy; anti-tumor chemotherapy in 6 months;
  2. lesions have been treated by irradiation;
  3. participate in other therapeutic or interventional clinical trials. - Page 5 of 5 [DRAFT] -
* Have central nervous system metastasis;
* History of other malignancies except carcinoma in-situ of uterine cervix, cured basal cell carcinoma of skin and other malignancies for more than 5 years;
* Have symptomatic ascites and need for treatment;
* Have serious concurrent illness including, but not limited to

  1. uncontrolled congestive heart failure(NYHA classification grade III or IV), unstable angina pectoris, unstable cardiac arrhythmias, uncontrolled moderate or serious hypertension(systolic blood pressure >21.3 Kpa or diastolic blood pressure >13.3 Kpa);
  2. ongoing or active serious infection;
  3. uncontrolled diabetes mellitus;
  4. psychiatric illness which potentially hamper the ability to willingly give written informed consent and compliance with the study protocol;
  5. HIV infection;
  6. other serious illness considered not suitable for this study by investigators.
* be allergic or have contraindications to target medicines involved in this study, gemcitabine or oxaliplatin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 1 year
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year. The progression is defined consistent with Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria for solid tumors.

SECONDARY OUTCOMES:
Overall survival | up to 2 years
Objective Response Rate | up to 1 year
  Objective Response Rate is defined as the percentage of patients with a complete or partial response to treatment, consistent with RECIST version 1.1 criteria for solid tumors.
Disease Control Rate | up to 1 year
  Disease Control Rate is defined as the percentage of patients with a complete or partial response to treatment or stable disease, consistent with RECIST version 1.1 criteria for solid tumors.
percentage of patients with Clinical Benefit Response | up to 1 year
  Composite measure based on patient-reported pain (per Faces pain scale revised), patient-reported pain medication, Karnofsky performance status(KPS), and weight. Clinical benefit is indicated by either:(a) improvement in pain (less pain intensity with stable or decreased pain medication; or less pain medication with stable or decreased pain intensity) with stable or improved KPS; or (b) improvement in KPS with stable or improved pain.With stable for KPS and pain, clinical benefit may be indicated with an observation of positive weight change.
  Clinical benefit response (CBR) was classified weekly and a patient was considered a clinical benefit responder if clinical benefit was observed and maintained over a 4 week period.

CONTACTS AND LOCATIONS:
Overall Officials: yingbin liu, PHD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided